CLINICAL TRIAL: NCT02614300
Title: The Role of Pulmonary Rehabilitation and Airways Clearance Techniques in the Multidisciplinary Management of Non CF Bronchiectasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Eva Polverino, Specialist in Respiratory Diseases, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: PulmRehab_NCFBE
Record Dates: First submitted 2015-11-18; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
Keywords: pulmonary rehabilitation; chest physiotherapy; non-cystic fibrosis bronchiectasis; exercise tolerance; bronchiectasis; respiratory therapy
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pulmonary Rehabilitation (Active Comparator): These sessions will be individually designed and they will be a combination of global aerobic interval training using a cycloergometer. The aim is to achieve a training intensity of 80% HR or greater of the obtained during the ISWT. This intensity will be progressively increased during the firsts four weeks until achieving the target. The duration will be of about 45 minutes per session. Oxygen Saturation, HR and Borg scale for dyspnoea and fatigue will be measured before, during and at the end of the session in order to monitories the effort.
  Interventions: Other: Pulmonary Rehabilitation
- Chest Physiotherapy (Active Comparator): The ELTGOL technique ("total slow expiration with glottis open in lateral decubitus") for airways clearance will be used in order to move respiratory secretions from the distal bronchial tree. It will be applied during 15 minutes each side (right and left lungs) assuming an approximate session length of 30 minutes. The patient could perform the cough technique when it's necessary.
  Interventions: Other: Chest Physiotherapy
- Pulmonary Rehabilitation and Chest Physiotherapy (Active Comparator): This group will perform a combination of the two programs in the same session with a total duration of 1h and 15 minutes. The session will be divided in different parts: First, we will execute 15min of chest physiotherapy (7.5min for each side); second, the pulmonary rehabilitation session (45min) and finally, another 15min of chest physiotherapy (7.5min for each side). The patient will have a rest when it's necessary and we will continue with the session when there is a decrease of 2 points in the Borg scale.
  Intensity of physiotherapy exercises and drainage techniques will be maintained similar to the PR and CP programs.
  Interventions: Other: Pulmonary Rehabilitation and Chest Physiotherapy
- Control Group (No Intervention): For the control group, participants will attend educational sessions to improve patients' understanding and awareness of the respiratory diseases. These sessions will be performed at beginning and at 12 weeks by the physiotherapist and the pulmonologist.
  The physiotherapist will also do monthly telephone calls for patient's monitoring.

INTERVENTIONS:
Other: Pulmonary Rehabilitation and Chest Physiotherapy — The patient will come 3 times per week during 12 weeks Each session 1h15min
  Arms: Pulmonary Rehabilitation and Chest Physiotherapy
Other: Pulmonary Rehabilitation — The patient will come 3 times per week during 12 weeks Each session 45min
  Arms: Pulmonary Rehabilitation
Other: Chest Physiotherapy — The patient will come 3 times per week during 12 weeks Each session 30min
  Arms: Chest Physiotherapy

SUMMARY:
Pulmonary rehabilitation programs are part of the multidisciplinary treatment of some chronic respiratory diseases such as COPD (chronic obstructive pulmonary disease). Although clinical guidelines of other diseases such as non-cystic fibrosis bronchiectasis (nCFBE) discuss the benefits of these programs in quality of life and exercise tolerance, evidence of such intervention in nCFBE patients is insufficient. Longer studies are needed with larger sample sizes and optimized to maximize the response and maintain long-term benefits. The present study aims to examine the effects in exercise tolerance of a pulmonary rehabilitation program combined with respiratory physiotherapy in patients with nCFBE. It is a randomized controlled clinical trial with a total duration of 24 months. The intervention will be performed during 12 weeks and then will be a period of 12 months of maintenance. This is a multicenter study involving the following Hospitals: Hospital Clinic, Hospital la Plató and Hospital del Mar of Barcelona, Hospital Josep Trueta of Girona, Royal Infirmary of Edinburgh and Fondazione Maugeri di Lumezzane of Italy. Subjects will be randomized into three groups in a ratio (1: 1: 1) (1) Pulmonary Rehabilitation (2) Chest Physiotherapy and (3) Pulmonary Rehabilitation + Chest Physiotherapy. Hospital la Plató from Barcelona will be responsible for carrying out the Control Group. The primary endpoint will be the test of "endurance shuttle walk test".

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50-80 years;
* No performing regular physiotherapy treatment or physical training (≤ 1 time/week);
* Stable disease [no changes in the chronic therapy (both inhaled and systematic) in the usual respiratory symptoms (according to the medical evaluation) and spirometry in the last 4 weeks prior to study recruitment];
* Regular cough and expectoration;
* Ability to follow the exercise program;
* Ability to perform all clinical tests, to understand the process and the purposes of the study;
* A history of at least 2 exacerbations during the previous year requiring antibiotic treatment and;
* Signed informed consent.

Exclusion Criteria:

* Active smokers, ex-smokers of less than 1 year prior to recruitment and/or a history of >20 smoking packs/year;
* FEV1 <30% or/and TLC<40% ;
* Diagnosis of cystic fibrosis, sarcoidosis, pulmonary fibrosis, active tuberculosis or non tuberculosis mycobacterial infection,
* Diagnosis of asthma or COPD as a primary respiratory disease and associated secondary bronchiectasis,
* Patients with unstable cardiac disease or locomotor difficulties that preclude exercise (eg, severe arthritis or severe peripheral vascular disease);
* Chronic respiratory failure and/or oxygen therapy;
* Frequent haemoptysis (≥ 2 times/month);
* Participation in a PR program during the year prior to inclusion or during the study protocol;
* Participation in a CP program during 1 month prior to inclusion;
* Any physical and psychological disorder that interferes with protocol compliance;
* Participation in a clinical trial implying any change in usual pharmacological treatment in the last 6 months before recruitment;
* Being on the waiting list for lung transplantation or have been transplanted.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Exercise tolerance capacity measured as the distance walked in meters during the shuttle test at constant speed (ESWT) at 12 weeks. | At Screening and 12 weeks of intervention

SECONDARY OUTCOMES:
Exacerbations incidence and symptoms | During all study (12 weeks of intervention)
Change from Baseline Health related quality of life at 12 weeks. | At Screening and 12 weeks of intervention with Quality of Life Questionnaire (QoL-B)
Change from Baseline Impact of expectoration on the quality of life at 12 weeks. | At Screening and 12 weeks of intervention with Leicester Cough Questionnaire (LCQ)
Sputum colour | During all study (12 weeks of intervention) with Murray's colour scale
Change from Baseline FEV1, FVC and FEV1/FVC at 12 weeks. | At Screening and 12 weeks of intervention with Pulmonary Function Tests
Change from Baseline Physical activity level measured by accelerometry at 12 weeks. | At Screening and 12 weeks of intervention with accelerometry
Sputum quantity | During all study (12 weeks of intervention) with weight of sputum containers in grams

REFERENCES:
- [Derived] Herrero-Cortina B, Alcaraz-Serrano V, Torres A, Polverino E. Reliability and Minimum Important Difference of Sputum Weight in Bronchiectasis. Respir Care. 2020 Oct;65(10):1478-1487. doi: 10.4187/respcare.07175. Epub 2020 Feb 18. PMID 32071136